CLINICAL TRIAL: NCT00005509
Title: Cardiovascular Risk Factors in a Cohort of Latina Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5027; R29HL059947 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To conduct a cross-sectional study of cardiovascular risk factors in a cohort of Latina women.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease (CVD) is the leading cause of death among Latina women (LW) in the United States. Nursing knowledge in the area of CVD and Latina women is currently underdeveloped. Most studies have included Mexican women with limited information on how predictors such as resources, situational, personal, and demographic factors have an effect on the CVD-related dietary practices, physical activity, and exercise practices among Latina women subgroups such as Central American women.

DESIGN NARRATIVE:

To conduct a cross-sectional and follow-up preliminary intervention study in order to describe and analyze the CVD-related diet, physical activity, and exercise practices predictors in 221 Mexican and Central American women recruited from six counties in Northern California. Face-to-face interviews were conducted with Mexican American and Central American women (ages 40-75) who had at least one risk factor for CVD to answer the following questions: What were the CVD-related risk factors, dietary practices, physical activity, and exercise behaviors in Mexican and Central American women who were 40 to 75 years and who had at least one risk factor for CVD? What was the relationship between predictor variables (resources, situational, personal, and demographic factors) with CVD-related diet practices, physical activity, and exercise behaviors (outcome variables)?, and what were the short and intermediate-term effects of a cardiovascular nursing intervention on diet, physical activity, and exercise? A sample of 221 women was targeted. Data were collected during the first two years of the project to provide substantial research-based information to develop a cardiovascular nursing intervention to support Latina women efforts to promote heart health and prevent CVD. Data were analyzed during the third year and the cardiovascular nursing intervention was developed to determine the short (3 months) and intermediate-term (6 months) effects in the outcome variables. A randomly selected sample of 60 women from the same cohort was randomly assigned to the developed intervention group (n=30 in each group) and to a delayed-intervention control group.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Juarbe — University of California, San Francisco

REFERENCES:
- [Background] Juarbe TC, Lipson JG, Turok X. Physical activity beliefs, behaviors, and cardiovascular fitness of Mexican immigrant women. J Transcult Nurs. 2003 Apr;14(2):108-16. doi: 10.1177/1043659602250623. PMID 12772619
- [Background] Juarbe T, Turok XP, Perez-Stable EJ. Perceived benefits and barriers to physical activity among older Latina women. West J Nurs Res. 2002 Dec;24(8):868-86. doi: 10.1177/019394502237699. PMID 12469724